CLINICAL TRIAL: NCT04615247
Title: A Feasibility Trial of a Group Based Yoga Intervention for Chronic Pelvic Pain in Women
Brief Title: Program to Overcome Pelvic Pain Study
Acronym: POPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Stanford University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-29762; R34AT010356 (NIH)
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pelvic Pain; Chronic Pelvic Pain; Recurrent Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Program (Experimental): The study yoga intervention is designed to provide instruction and practice in selected yoga postures and techniques chosen by an expert panel for their potential to improve pelvic pain in women.
  Interventions: Other: Yoga Program
- Physical Conditioning Program (Active Comparator): A low-impact, muscle stretching and strengthening program.
  Interventions: Other: Physical Conditioning Program

INTERVENTIONS:
Other: Yoga Program — The yoga program is designed to maximize women's awareness of and control over the pelvic floor, promote relaxation, and improve physical function.
  Arms: Yoga Program
Other: Physical Conditioning Program — The physical conditioning program will focus on a core set of exercises designed to improve physical function and emotional well-being in order to improve management of chronic pain.
  Arms: Physical Conditioning Program

SUMMARY:
To refine and evaluate the feasibility of procedures for a future full-scale efficacy trial of a group-based therapeutic yoga intervention versus physical conditioning (stretching and strengthening) intervention for women with chronic pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older who report chronic or recurrent pelvic pain for at least 6 months
* Report an average daily pain intensity score of at least 4 (on a 0 to 10 scale) on a screening 7-day pain log
* Report prior clinical evaluation of pain by a healthcare professional including at least a superficial pelvic exam
* Willing to refrain from initiating new clinical treatments that may affect their pain during the study period

Exclusion Criteria:

* Report pelvic pain occurring exclusively with menses or exclusively during sexual intercourse (note that women with at least some pain between menses or intercourse are still eligible)
* Participation in organized yoga classes or muscle strengthening programs (e.g., Pilates) in the past month, or prior yoga therapy specifically directed a pelvic pain
* Currently pregnant (by self-report or screening test), pregnant within the past 6 months, or planning pregnancy
* Diagnosed with an alternate, reversible cause of pain that is unlikely to respond to yoga and requires another treatment modality (e.g., current pelvic infection or a gynecologic dermatosis)
* Initiation, dose escalation, or weaning of pharmacologic agents that may affect pelvic pain severity in the past 1 month (e.g., pain medications, antidepressants, anticonvulsants)-note that women on stable doses will be eligible
* Surgery to the genital or pelvic structures within 3 months, or prior cancer or irradiation to these structures
* Use of formal psychological therapies specifically for pelvic pain (e.g., systematic desensitization, sex therapy, cognitive therapy, relaxation therapy) within 1 month of screening
* Use of formal behavioral therapies for pelvic or genital pain (e.g., pelvic floor rehabilitation or biofeedback performed by a certified healthcare practitioner) within 1 month of screening
* Unable to walk up a flight of stairs or at least 2 blocks on level ground (i.e., functional capacity < 4 METs), or unable to get up from a supine to a standing position without assistance
* Participation in another interventional study that might interfere with or confound study procedures
* Known conflict with multiple available intervention class dates
* Inability to sign an informed consent or fill out questionnaires or complete study interviews in English, or lacking technical requirements to complete intervention classes or study visits by video

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Huang, MD, MAS, MPhil, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Yes
Starting no later than 6 months following publication of the main trial results (including on-line publication), the investigative team will make publically available de-identified individual participant data that underlie the results reported in the publication. This will include data about the baseline characteristics of the study participants and any primary or secondary trial outcomes presented in the publication.
Supporting Information: Study Protocol, ICF
Access Criteria: To gain access, data requestors will be asked to sign a data access agreement. In addition to signing a data access agreement, data requestors seeking to use trial data to generate new publications or presentations will be asked to submit a publication/presentation proposal that will be reviewed by the members of the trial steering committee, made up of the principal and co-investigators, for overlap with existing publication/presentation proposals as well as methodological appropriateness.

REFERENCES:
- [Derived] Huang AJ, Subak LL, Rowen TS, Schembri M, Raghunathan H, Gibson C, Pawlowsky S, Cheng J, Chao MT. A Multisite Randomized Feasibility Trial of a Remotely Delivered Pelvic Yoga Program for Women with Chronic Pelvic Pain Syndrome. J Integr Complement Med. 2025 May;31(5):483-492. doi: 10.1089/jicm.2024.0682. Epub 2024 Dec 26. PMID 39723995

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga Program | Physical Conditioning Program
Started | 17 | 19
Completed | 16 | 16
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Program | Physical Conditioning Program | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (15.4) | 52.4 (12.7) | 51.0 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 16 | 28
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Randomized Participants Who: a) Are Retained at 8 Weeks, b) Attend at Least 75% of Intervention Classes, c) Demonstrate at Least Moderate Intervention Self-efficacy, and d) Provide Pain Outcomes Data at 8 Weeks.
Description: Number of randomized participants who: a) are retained at 8 weeks, b) attend at least 75% of intervention classes, c) demonstrate at least moderate intervention self-efficacy, and d) provide pain outcomes data at 8 weeks.
Time Frame: 8 weeks
Population: Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 17 | 19
Participants | 14 | 12

2. Secondary Outcome: Percentage of Screenees Who Are Eventually Randomized
Description: Percentage of screenees who are eventually randomized
Time Frame: Randomization
Population: Screened Individuals
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 17 | 19
Participants | 17 | 19

3. Secondary Outcome: Percentage of Randomized Participants Who Drop Out by 8 Weeks
Description: Percentage of randomized participants who drop out by 8 weeks
Time Frame: 8 weeks
Population: Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 17 | 19
Participants | 1 | 3

4. Secondary Outcome: Percentage of Non-drop-outs Completing at Least 75% of Intervention Classes Over 8 Weeks
Description: Percentage of non-drop-outs completing at least 75% of intervention classes over 8 weeks
Time Frame: 8 weeks
Population: Randomized Participants who did not drop out
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 16 | 16
Participants | 15 | 13

5. Secondary Outcome: Percentage of Non-drop-outs Completing at Least 75% of Home Intervention Practice Over 8 Weeks
Description: Percentage of non-drop-outs completing at least 75% of home intervention practice over 8 weeks
Time Frame: 8 weeks
Population: Randomized Participants who did not drop out
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 16 | 16
Participants | 14 | 12

6. Secondary Outcome: Percentage of Participants With at Least Moderate Self-efficacy in Performing Postures/Exercises at 8 Weeks
Description: Participants will rate their self-confidence in performing each posture/exercise on a 5-point Likert scale (5-extremely, 4-very, 3-moderately, 2-somewhat, and 1-not at all confident. The percentage of participants with an average self-confidence score of 3 or higher across postures/exercises at 8 weeks will be calculated.
Time Frame: 8 weeks
Population: Randomized Participants who Submitted Self-Efficacy Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 15 | 16
Participants | 15 | 14

7. Secondary Outcome: Percentage of Participants Rated by a Consultant as Being at Least Moderately Competent in Performing Postures/Exercises at 8 Weeks
Description: Expert consultants will observe and rate participants' success in performing each posture/exercise on a 5-point Likert scale (5-extremely, 4-very, 3-moderately, 2-somewhat, and 1-not at all confident. The percentage of participants with an average competence rating of 3 or higher across postures/exercises at 8 weeks will be calculated.
Time Frame: 8 weeks
Population: Randomized Participants who Evaluated by Consultant
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 15 | 12
Participants | 15 | 12

8. Secondary Outcome: Percentage of Participants With Expected Pain Logs Returned at 8 Weeks
Description: Percentage of participants with expected pain logs returned at 8 weeks
Time Frame: 8 weeks
Population: Randomized Participants who did not drop out
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 16 | 16
Participants | 15 | 15

9. Secondary Outcome: Percentage of Participants With Expected Pain Interference Questionnaires Returned at 8 Weeks
Description: Percentage of participants with expected pain interference questionnaires returned at 8 weeks
Time Frame: 8 weeks
Population: Randomized Participants who did not drop out
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 16 | 16
Participants | 14 | 15

10. Secondary Outcome: Percentage of Participants With Expected Pelvic Pain Impact Measures Returned at 8 Weeks
Description: Percentage of participants with expected pelvic pain impact measures returned at 8 weeks
Time Frame: 8 weeks
Population: Randomized Participants who did not drop out
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Program | Physical Conditioning Program
Number analyzed (Participants) | 16 | 16
Participants | 14 | 15

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Yoga Program | Physical Conditioning Program
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 14/17 | 17/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Program (N=17) | Physical Conditioning Program (N=19)
Abdominal Pain Aggravated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallstones (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cold (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 1 (1)
Ebv Infection (Infections and infestations) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Knee Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thigh Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination Adverse Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Wrist Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Cystitis Interstitial (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic Pain Female (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Carpal Tunnel Release (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT04615247/Prot_SAP_000.pdf